CLINICAL TRIAL: NCT02547987
Title: CADENCE: Carboplatin and Docetaxel in Neoadjuvant Treatment of ER-Negative, HER2-Negative Breast Cancer: A Co-Clinical Trial With Genoproteomic Discovery
Brief Title: Neoadjuvant Carboplatin and Docetaxel in Triple Negative Breast Cancer
Acronym: CADENCE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mothaffar Rimawi (Other)
Responsible Party: Sponsor-Investigator, Mothaffar Rimawi, Associate Professor, Baylor Breast Care Center
Organization: Baylor Breast Care Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H- 36960 CADENCE
Record Dates: First submitted 2015-09-10; First posted 2015-09-14 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; triple negative; TNBC; triple negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel/Carboplatin (Experimental): Docetaxel 75 mg/m2 plus Carboplatin AUC 6 IV on Day 1 of each 21 day cycle for 6 cycles
  Interventions: Drug: Docetaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/m2 intravenously on day 1 of each 21-day cycle. Number of Cycles: 6
  Other Names: Taxotere
Drug: Carboplatin — Carboplatin AUC 6 intravenously on day 1 of each 21-day cycle. Number of Cycles: 6
  Other Names: Paraplatin

SUMMARY:
The purpose of this study is to determine whether the combination of docetaxel and carboplatin is an effective treatment for patients with triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To determine whether neoadjuvant docetaxel and carboplatin will increase the pCR rate in TNBC compared to historical controls. Pathologic complete response (pCR) will be defined as no residual invasive breast cancer in the breast and ipsilateral axillary lymph node (ypT0-is ypN0).

ELIGIBILITY:
Inclusion Criteria:

* All patients must be 18 years of age or older.
* All patients must be diagnosed with invasive breast cancer.
* Breast cancer must be ER-negative, and HER-2 negative according to CAP/ASCO biomarkers testing guidelines. Tumors may be PgR positive with an Allred score of less than 5.
* Primary breast tumor size at least 2 cm in one dimension by clinical or radiographic exam. Patients who have multicentric breast cancer are eligible if each lesion is estrogen receptor negative and HER2-negative. In that case, one lesion needs to be identified as the index lesion to be followed for clinical response. The index lesion must also be the lesion from which core biopsies are obtained.
* Patients with inflammatory breast cancer are eligible if they meet both of the following criteria:

  1. Patient has an underlying, clinically palpable breast mass of at least 2cm, AND
  2. a corresponding lesion is visualized on mammogram or ultrasound
* Normal bone marrow and organ function as defined below:

  * Leukocytes > 3,000/mcL
  * Absolute neutrophil count > 1,200/mcl
  * Platelets > 100,000/mcl
  * Serum bilirubin ≤ institutional 1.5 times upper limit of normal (ULN)
  * Aspartate aminotransferase/alanine aminotransferase ≤ 2.5 times ULN
  * Creatinine ≤ 1.5 ULN
* Women of childbearing potential (defined as women under the age of 55 with intact ovaries and uterus) must agree to use adequate contraception prior to study entry and for the duration of study participation. They must also have a negative urine pregnancy test within 7 days of starting treatment.
* Ability to understand and willingness to sign an IRB approved written informed consent document and follow study procedures including willingness to undergo study biopsies.

Exclusion Criteria:

* Any prior systemic therapy for breast cancer within 5 years.
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Patients with known bilateral invasive breast cancer. Patients with contralateral in situ breast carcinoma are eligible.
* Inflammatory breast cancer.
* Patients with confirmed stage IV disease.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxel or carboplatin.
* Known to be seropositive for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* If the patient is otherwise not deemed a good study candidate by sole discretion of the principal investigator.
* Patient is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2025-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - TriHealth Hatton Research, Cincinnati, Ohio
  - Lester & Sue Smith Breast Center at Baylor College of Medicine, Houston, Texas
  - Harris Health System Smith Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ademuyiwa FO, Chen I, Luo J, Rimawi MF, Hagemann IS, Fisk B, Jeffers G, Skidmore ZL, Basu A, Richters M, Ma CX, Weilbaecher K, Davis J, Suresh R, Peterson LL, Bose R, Bagegni N, Rigden CE, Frith A, Rearden TP, Hernandez-Aya LF, Roshal A, Clifton K, Opyrchal M, Akintola-Ogunremi O, Lee BH, Ferrando-Martinez S, Church SE, Anurag M, Ellis MJ, Gao F, Gillanders W, Griffith OL, Griffith M. Immunogenomic profiling and pathological response results from a clinical trial of docetaxel and carboplatin in triple-negative breast cancer. Breast Cancer Res Treat. 2021 Aug;189(1):187-202. doi: 10.1007/s10549-021-06307-3. Epub 2021 Jun 26. PMID 34173924

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patient eligibility is confirmed by both the study coordinator and a Lester & Sue Smith Breast Center physician. If a patient does not meet an inclusion criterion, or meets an exclusion criterion, as listed in the protocol section, the patient is excluded.
Groups:
- Docetaxel/Carboplatin: Docetaxel 75 mg/m2 plus Carboplatin AUC 6 IV on Day 1 of each 21 day cycle for 6 cycles
  Docetaxel/Carboplatin: Docetaxel 75 mg/m2 plus Carboplatin AUC 6 IV (in the vein) on day 1 of each 21-day cycle. Number of Cycles: 6
Period: Overall Study
Arm/Group | Docetaxel/Carboplatin
Started | 25
Completed | 22
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel/Carboplatin
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response
Description: This is the complete disappearance of invasive cancer in the breast at the time of surgery
Time Frame: At the time of definitive surgery (approximately 4-5 months after beginning chemotherapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel/Carboplatin
Number analyzed (Participants) | 25
Participants | 10

ADVERSE EVENTS:
Time Frame: 6.5 months (from screening/baseline to 30 days after completion of all cycles).
Description: Adverse events were assessed at baseline, at the start of each 21-day cycle, and up to 30 days after completion of all cycles using descriptions and grading scales found in CTCAE v4.0.
Arm/Group | Docetaxel/Carboplatin
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 3/25
Other Adverse Events (participants affected / at risk) | 16/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel/Carboplatin (N=25)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel/Carboplatin (N=25)
Anemia (Blood and lymphatic system disorders) | 9 (15)
Eyelid function disorder (Eye disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 7 (15)
Dyspepsia (Gastrointestinal disorders) | 4 (5)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (7)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 8 (13)
Pain (General disorders) | 2 (2)
Skin infection (Infections and infestations) | 3 (4)
Alanine aminotransferase increased (Investigations) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 4 (5)
Creatinine increased (Investigations) | 2 (3)
Lymphocyte count decreased (Investigations) | 3 (7)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 6 (9)
White blood cell decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (7)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 6 (6)
Headache (Nervous system disorders) | 5 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4)
Insomnia (Psychiatric disorders) | 3 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (11)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT02547987/Prot_SAP_000.pdf